CLINICAL TRIAL: NCT03019783
Title: Atazanavir and Endothelial Function in Older HIV Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua A. Beckman, MD, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AI424-469
Record Dates: First submitted 2016-12-08; First posted 2017-01-13 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: HIV
Keywords: Endothelial function
MeSH Terms: interventions — Atazanavir Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remains on baseline HIV regimen (Placebo Comparator): Subjects are enrolled and either kept on their baseline regimen. This is being designated the placebo comparator.
  Interventions: Other: Placebo
- Atazanavir switch (Active Comparator): These subjects are switched to an atazanavir-based regimen.
  Interventions: Drug: Atazanavir

INTERVENTIONS:
Drug: Atazanavir — The active group will switch from a non-atazanavir regimen to an atazanavir-based regimen.
  Other Names: Reyataz
  Arms: Atazanavir switch
Other: Placebo — The control group will stay on their baseline regimen
  Arms: Remains on baseline HIV regimen

SUMMARY:
The investigators hypothesize that older subjects with HIV randomly assigned to atazanavir will have increased bilirubin levels, reduced oxidative stress, and improved flow-mediated, endothelium-dependent vasodilation compared to subjects not switched to atazanavir.

DETAILED DESCRIPTION:
The mortality induced by HIV has dropped significantly due to effective antiretroviral therapy. Epidemiological data suggest a less than 5% 10-year mortality for patients treated with HAART. As a result of the reduction in early AIDS-related deaths, HIV has become a chronic disease manifesting the common components of chronic disease such as inflammation, vascular dysfunction, and oxidative stress. The combination of these trends put HIV patients at increased risk of myocardial infarction compared with age-matched subjects over the long term. Several studies suggest that some protease inhibitors might increase the risk of myocardial infarction. The leading theory behind this association derives from the relationship between protease inhibitor use and the onset of an atherogenic dysmetabolism including the development of insulin resistance, dyslipidemia, and oxidative stress.

In contrast to the older protease inhibitors, atazanavir induces neither insulin resistance nor dyslipidemia. In addition, atazanavir has a property unique among protease inhibitors: elevation of unconjugated bilirubin by inhibiting the enzyme uridine diphosphate glucuronyltransferase (UGT) 1A1. Bilirubin is a potent intracellular antioxidant. The investigators have demonstrated that higher levels of bilirubin within the normal range are associated with reduced rates of stroke and peripheral artery disease. Patients with Gilbert's Syndrome (chronic elevations of bilirubin as a result of genetically reduced UGT 1A1) have a lower rate of myocardial infarction compared with age-matched controls. It is plausible that use of atazanavir compared with other protease inhibitors, by reducing oxidative stress, may improve vascular function and, ultimately, reduce the rate of cardiovascular complications with chronic therapy.

The benefit of atazanavir may be particularly important now with the aging of the HIV population. Aging is associated with higher levels of oxidative stress and endothelial dysfunction, both of which are associated with heightened rates of cardiovascular morbidity and mortality. Accordingly, the investigators hypothesize that the use of atazanavir in stable HIV patients age 45 years or older will improve endothelial dysfunction and reduce oxidative stress compared with continuing the current therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Stable non-atazanavir-containing regimen consisting of co-formulated tenofovir/emtricitabine as the NRTIs plus a third agent for 3 months or longer. The third agent can be any FDA-approved PI, NNRTI, or raltegravir.
* HIV RNA < 200 cop/mL at screening and at least once within the prior year,
* No treatment interruptions > 7 days in the 3 months prior to study entry
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Signed Written Informed Consent. Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug to minimize the risk of pregnancy.
* WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

  * Amenorrhea that has lasted for 12 consecutive months without another cause, or
  * For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
  * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.
  * WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of the investigational product.

Exclusion Criteria:

* Sex and Reproductive Status

  * WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the last dose of study drug.
  * Women who are pregnant or breastfeeding.
  * Women with a positive pregnancy test.
* Target Disease Exceptions

  * Prior treatment failure on or intolerance to atazanavir
  * Known or suspected resistance to atazanavir
  * Receiving ART different from co-formulated tenofovir/emtricitabine plus third agent (PI, NNRTI, or raltegravir) regimen
  * Receiving Viagra, Levitra, or Cialis
  * A new AIDS-defining condition diagnosed within the 30 days prior to screening
  * Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Medical History and Concurrent Diseases

  * Patients with Gilbert's Syndrome or elevated bilirubin levels (>1.5 mg/dL) at baseline (for the randomized trial)
  * Patients with uncontrolled diabetes (hemoglobin A1c > 11%)
  * Patients allergic to nitroglycerin
* Prohibited Treatments and/or Therapies

  * Recent initiation of hormones or immunomodulators (3 months)
  * Current receipt of proton-pump inhibitor therapy
* Other Exclusion Criteria

  * Prisoners, or subjects who are involuntarily incarcerated.
  * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
  * Subjects for whom the investigators believe there will be a low likelihood of medication compliance.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Beckman, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beckman JA, Wood BR, Ard KL, Price CN, Solomon DA, Zuflacht JP, Milian J, Prenner JC, Sax PE. Conflicting effects of atazanavir therapy on atherosclerotic risk factors in stable HIV patients: A randomized trial of regimen switch to atazanavir. PLoS One. 2017 Oct 12;12(10):e0181993. doi: 10.1371/journal.pone.0181993. eCollection 2017. PMID 29023508

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remains on Baseline HIV Regimen | Atazanavir Switch
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remains on Baseline HIV Regimen | Atazanavir Switch | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6) | 53 (6) | 53 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 23 | 18 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 18 | 30
  White | 17 | 13 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated, Endothelium-dependent Vasodilation
Description: The investigators will evaluate flow-mediated, brachial artery vasodilation (percentage increase in diameter in response to a 5 minute ischemic challenge) at study entry and then after 28 days, with the change between the two measurements being the primary endpoint.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage vasodilation
Arm/Group | Remains on Baseline HIV Regimen | Atazanavir Switch
Number analyzed (Participants) | 29 | 31
percentage vasodilation | 0.2 (2.4) | 0.8 (4.6)

2. Secondary Outcome: Change in Plasma Total Antioxidant Capacity
Description: The investigators will evaluate plasma total antioxidant capacity at study entry and then after 28 days, with the change between the two measurements being the secondary endpoint.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Remains on Baseline HIV Regimen | Atazanavir Switch
Number analyzed (Participants) | 29 | 31
micromolar | -21 (271) | 219 (213)

ADVERSE EVENTS:
Time Frame: 1 month
Description: No adverse events
Arm/Group | Remains on Baseline HIV Regimen | Atazanavir Switch
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

LIMITATIONS AND CAVEATS:
There were no limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No